CLINICAL TRIAL: NCT01353092
Title: PEMF Treatment in Patients With Treatment Resistant Depression in On-going Antidepressant Drug Therapy. A Randomized, Double-blind, Clinically Controlled, Dose-response PEMF Trial for a Duration of Eight Weeks
Brief Title: Pulsating ElectroMagnetive Treatment (PEMF) at Treatment Resistant Depression
Acronym: PEMFII
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hillerod Hospital, Denmark (Other)
Responsible Party: Principal Investigator, Per Bech, Professor, Hillerod Hospital, Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 26.04.2010
Record Dates: First submitted 2011-04-27; First posted 2011-05-12 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Treatment Resistant Depression
Keywords: Randomized Controlled Trial; Major depression; Hamilton; PEMF
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active PEMF twice daily (Experimental): Re5 treatment helmet using Pulsating ElectroMagnetic Field:
  Intervention: 30 minutes of active PEMF therapy in the morning and 30 minutes of active PEMF therapy in the afternoon
  Interventions: Device: Re5 Pulsating ElectroMagnetic Fields
- Active PEMF once daily (Active Comparator): Re5 treatment helmet using Pulsating ElectroMagnetic Field:
  Intervention: 30 minutes of sham therapy and 30 minutes of active therapy (morning or afternoon)
  Interventions: Device: Re5 Pulsating ElectroMagnetic Fields (PEMF)

INTERVENTIONS:
Device: Re5 Pulsating ElectroMagnetic Fields — Re5 Treatment Helmet using Pulsating ElectroMagnetic Fields (PEMF):
  30 minutes of active PEMF therapy in the morning and 30 minutes of active PEMF therapy in the afternoon
  Other Names: T-PEMF = Transcranially applied PEMF
  Arms: Active PEMF twice daily
Device: Re5 Pulsating ElectroMagnetic Fields (PEMF) — Re5 Treatment Helmet using Pulsating ElectroMagnetic Fields (PEMF):
  30 minutes of sham therapy and 30 minutes of active therapy (morning or afternoon)
  Other Names: T-PEMF = Transcranially applied PEMF
  Arms: Active PEMF once daily

SUMMARY:
In this study patients with treatment resistant depression, as defined by Harold Sackeim, is subjected to daily sessions, for eight weeks, with Pulsating ElectroMagnetive Treatment (PEMF). Treatment is given two times a day, in the morning and in the afternoon. Patients are randomized into two groups. In group A patients receive active treatment both morning and afternoon. In group B patients receive one sham and one active treatment. The study is double-blind as neither the assessors or patients are aware of treatment allocation. Each session lasts 30 minutes. Patients are psychometrically assessed weekly for depression severity and side effect. After this intervention period patients are followed for further three weeks without PEMF treatment. Patients are on unchanged medication for the whole of the study period.

ELIGIBILITY:
Inclusion Criteria:

* Treatment resistant Major depression (grade 3 Sackeim criteria)
* Age above 18 and below 85
* Hamilton (17 item version) score above 12
* Unchanged psychopharmacological treatment for last five weeks.

Exclusion Criteria:

* suicidality above 2 on item three on Hamilton scale or,earlier PEMF treatment
* dementia or similar cognitive impairment
* psychotic disorder
* abuse of alcohol or drugs
* pregnant or lactating women
* insufficient birth control measures

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2011-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Hamilton depression rating scale | Every week for 11 weeks
  Interviewer based rating scale to measure severity of depression

SECONDARY OUTCOMES:
UKU | Every week for 11 weeks
  Side effect scale

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Lunde, Coordinator, Principal Investigator — Mental Health Centre North Zealand Psychiatric Research Unit
Locations (1):
- Psychiatric Research Unit, Mental Health Centre North Zealand, Hilleroed, Denmark

REFERENCES:
- [Background] Martiny K, Lunde M, Bech P. Transcranial low voltage pulsed electromagnetic fields in patients with treatment-resistant depression. Biol Psychiatry. 2010 Jul 15;68(2):163-9. doi: 10.1016/j.biopsych.2010.02.017. Epub 2010 Apr 10. PMID 20385376
- [Derived] Bech P, Timmerby N, Martiny K, Lunde M, Soendergaard S. Psychometric evaluation of the Major Depression Inventory (MDI) as depression severity scale using the LEAD (Longitudinal Expert Assessment of All Data) as index of validity. BMC Psychiatry. 2015 Aug 5;15:190. doi: 10.1186/s12888-015-0529-3. PMID 26242577